CLINICAL TRIAL: NCT01374932
Title: The CPASMA Trial: Is There an Improvement in Asthma in Patients With Both Asthma and Obstructive Sleep Apnoea Syndrome (OSAS) Treated With Continuous Positive Airway Pressure (CPAP) After Six Months?
Brief Title: CPASMA: Is There an Improvement in Asthma in Patients With Both Asthma and OSAS Treated With CPAP?
Acronym: CPASMA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cimera (Network)
Responsible Party: Principal Investigator, Dr. Joan B Soriano, Programme Director, Cimera
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The CPASMA trial
Record Dates: First submitted 2011-05-30; First posted 2011-06-16 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Asthma; Obstructive Sleep Apnea Syndrome
Keywords: Asthma; Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Asthma; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPAP (see below) (Experimental): Adult patients with asthma who require treatment with CPAP because of OSAS (RDI> = 20 events per hour). CPAP will be administered according to SEPAR guidelines and tailored to individual characteristics
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — Continuous positive airways pressure (CPAP)
  Other Names: Brand names will be added during fieldwork

SUMMARY:
The CPASMA trial is a descriptive, prospective, multicentre clinical trial, with a before/after Continuous Positive Airway Pressure (CPAP) assessment in participating patients. It aims to answer the following question: Is there an improvement in asthma in those patients with both asthma and obstructive sleep apnoea syndrome (OSAS) treated with CPAP after six months?. It is hypothesized that treatment of OSAS with CPAP in patients with both OSAS and asthma concommitantly, may have a beneficial effect also on asthma outcomes. This clinical effect in asthma could be assessed objectively by applying validated questionnaires for quality of life and asthma control.

DETAILED DESCRIPTION:
Full protocol in Spanish, available upon request

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 to 70 yrs.) with asthma who require treatment with CPAP because of OSAS (RDI> = 20 events per hour)

Exclusion Criteria:

* unstable or severe comorbidity,
* patients in treatment with drugs that interfere with the clinical course of asthma and/or OSAS,
* cognitive/psychiatric disorders that preclude patient participation/cooperation,
* COPD or other lung disease accompanied by chronic airflow limitation, and
* any clinical condition considered severe enough by the investigators to preclude all the diagnostic and therapeutic procedures outlined in this protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Asthma control questionnaire | 6 months
  Changes in clinical and functional variables and in the asthma control questionnaire (ACQ) in the period prior to start the CPAP treatment and after a 6-months follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Jose Serrano, MD, Principal Investigator — Hospital de Inca
Locations (10):
- Spain (10):
  - Hospital comarcal de Inca, Inca, Balearic Islands
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital de Jerez, Cadiz
  - Hospital de Laredo, Cantabria.
  - Hospital Universitario Dr. Negrín, Las Palmas
  - Hospital Moncloa, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Corporació Sanitària Parc Taulí, Sabadell